CLINICAL TRIAL: NCT06195748
Title: The Effect of Ankle Kinesio Taping on Balance and Functional Performance in Obese Female Collegiate Students
Brief Title: Ankle Kinesio Taping on Balance and Functional Performance in Obese Females.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Morgan Allam, Assistant Professor of physical therapy for surgery, Faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB Approval No. 2023-124
Record Dates: First submitted 2023-12-23; First posted 2024-01-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Kinesiotape Group) (Experimental): The technique will follow manufacturer's guidelines, which is described in the Kinesio taping method. According to the manufacturer, the controllable variables in KT application included degree of pre-stretch applied to the tape (75-100%), the location and treatment goals. The subject will be asked to lie supine, with the ankle of the dominant side in neutral position. A Y shaped KT strip will be applied from the heel to lateral and medial femoral condyles. A I shaped KT strip will be applied from medial malleolus to lateral malleolus, passing under the heel. Another I shaped KT strip will be applied from slightly above the medial malleolus to slightly above the lateral malleolus, crossing on the instep at the malleoli level.
  Interventions: Other: Kinesiotaping
- Group B (Placebo KT Group) (Placebo Comparator): The same tape will be used for the interventional application. Two strips will be used, one from the heel to the proximal third of the leg, the other from the lateral malleolus to the medial malleolus crossing on the instep, both with 0 tension
  Interventions: Other: Placebo kinesiotaping

INTERVENTIONS:
Other: Kinesiotaping — According to the manufacturer, the controllable variables in KT application included degree of pre-stretch applied to the tape (75-100%), the location and treatment goals. The subject will be asked to lie supine, with the ankle of the dominant side in neutral position. A Y shaped KT strip will be applied from the heel to lateral and medial femoral condyles. A I shaped KT strip will be applied from medial malleolus to lateral malleolus, passing under the heel. Another I shaped KT strip will be applied from slightly above the medial malleolus to slightly above the lateral malleolus, crossing on the instep at the malleoli level.
  Arms: Group A (Kinesiotape Group)
Other: Placebo kinesiotaping — The same tape will be used for the interventional application with 0 tension.
  Arms: Group B (Placebo KT Group)

SUMMARY:
Obesity is one of the most dangerous factors affecting the joints, which must be prevented due to arthritis and the long-lasting, tiring effects that affect a person's life [1], The most important of these are foot problems due to weight and excess pressure, It is also one of the factors that greatly affects walking movement because it increases the load on joint movement, This increases the risk of musculoskeletal diseases.

DETAILED DESCRIPTION:
It had been reported that obese subjects have a higher prevalence of falls and ambulatory stumbling or a loss of balance than their non-obese counterparts. Excess weight increases the stress within the bones, joints, and soft tissues, resulting in impaired musculoskeletal function. such as abnormal mechanics of the body. These impairments, such as impaired balance, gait, strength, sensory function, and neuromuscular function have been identified as strong risk factors for falls.

Participants that are eligible to participate to the study will be distributed into two groups: Group A will receive ankle kinesiotaping on the dominant leg. While, Group B will receive placebo kinesiotaping on the dominant leg. The treatment duration will be 6 weeks for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Female students between 18 and 25 years old
* BMI of 30 kg/ m2 or more

Exclusion Criteria:

* Orthopedic or neurosurgery injury past 6 months
* Ankle edema
* Skin allergy to the tape
* Abnormalities of the nervous system
* Any previous history of injury
* Use of medication in the past 3 months
* Regular physical activity at least three times a week

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Static balance | 6 weeks
  Single leg stance test: It is used for assessment of static balance. The participants will be instructed to close their eyes, stand barefoot on the dominate and then on non-dominant leg, and elevate the other limb so that it is close to but not touching the ankle of the limb on which they are stanced. The individual will be told to cross her arms over her chest before lifting the limb. The length of time the person can stand on one leg will be timed by the investigator using a stopwatch.

SECONDARY OUTCOMES:
Dynamic balance | 6 weeks
  the Biodex Balance System (BBS) SD (12.1-inch [30.7-cm] display, 115 VAC; Biodex Medical Systems Inc., Shirley, NY, USA). The BBS measures stability indices, which represent the variance of foot platform displacement in degrees for motion in different planes. The platform is fixable and movable.
Single leg hop test | 6 weeks
  The students will be asked to perform a maximum forward jump and land on the tested leg (first with the dominant, then with the non-dominant) while maintaining a two-second landing posture. The distance between the rear foot at landing and the start point will be measured in centimeter after being normalized to the subject leg length. The test result will be calculated as the average of the two best performances out of three trials
Single leg vertical jump | 6 weeks
  The students will be advised to stand on one leg, approximately one foot from the wall, and use the index finger to mark the wall as a reference point. Then they will jump on one leg (the dominant) three times and then the other leg (the non-dominant) three times. The difference between these two points was determined in centimeter, and the test result will be recorded as an average.

CONTACTS AND LOCATIONS:
Overall Officials: Hadaya M Eladl, PhD, Study Director — Assisstant professor of physical therapy for surgery, Faculty of physical therapy
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allam NM, Eladl HM, Elsherbini DMA, Abulfaraj M, Almadani ME, Megahed Ibrahim A, El-Sherbiny M, Eladl MA, Nosseir N, Jamjoom R. Efficacy of ankle Kinesio taping on balance and functional performance in obese female collegiate students: a prospective randomized placebo-controlled trial. Front Public Health. 2025 Aug 11;13:1631757. doi: 10.3389/fpubh.2025.1631757. eCollection 2025. PMID 40860562